CLINICAL TRIAL: NCT06399705
Title: REvascularization CHoices Among Under-Represented Groups Evaluation: The RECHARGE Trial - Minorities
Acronym: RECHARGE:M
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-11026800 - 2
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease
Keywords: RECHARGE; Cardiac Surgery; Minority; percutaneous coronary intervention; Quality of Life
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass; Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The researchers and most study personnel (including those from the QOL follow-up center and events assessors, clinical events committee and angiographic core laboratory) will be blinded to allocated treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RECHARGE: Minorities - CABG (Other)
  Interventions: Procedure: Coronary artery bypass grafting
- RECHARGE: Minorities - PCI (Other)
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Coronary artery bypass grafting — Coronary artery bypass grafting (CABG), also called heart bypass surgery, is a medical procedure to improve blood flow to the heart.
  Other Names: CABG
  Arms: RECHARGE: Minorities - CABG
Procedure: Percutaneous coronary intervention — Percutaneous coronary intervention (PCI) is a non-surgical procedure used to treat the blockages in a coronary artery; it opens up narrowed or blocked sections of the artery, restoring blood flow to the heart
  Other Names: PCI
  Arms: RECHARGE: Minorities - PCI

SUMMARY:
This is a research study in minorities to compare the outcomes of two procedures that restore blood flow to the arteries of the heart. In one procedure the blockages are ballooned and then stented with a small wire mesh tube through a small incision in the wrist or the groin. The other procedure is an open-heart operation in which healthy blood vessels from inside the chest, leg, and/or forearm are used to "bypass" the blockages (like a detour). Outcomes will be measured by comparing survival and improvement in quality-of-life.

DETAILED DESCRIPTION:
The RECHARGE: Minorities Trial is a multicenter, 1:1 randomized, open-label superiority trial.

Patients meeting the eligibility criteria for whom there is equipoise for revascularization with CABG and PCI, as determined by the local Heart Team, will be included. Participants will be followed for 5-10 years. Telephone follow-up will be conducted by the a central follow-up coordinating center at 30 days, 3 months, 6 months, and thereafter every 6 months through 36 months post-randomization. After 36 months, follow-up will be performed every year (48, 60, 72, 84, 96, 108, 120 months). A repeat transthoracic echocardiogram and blood draw for serum creatinine, hemoglobin and lipids should be performed at 1 year, as per standard of care, at either an out-patient facility or in a hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must identify as a minority
2. Patient is at least 18 years old.
3. Multivessel or left main CAD is present for which revascularization is intended and for which there is equipoise between CABG and PCI according to local Heart Team assessment.
4. Ability to provide written informed consent and comply with all follow-up procedures, including QOL questionnaires.

Exclusion Criteria:

1. ST-segment elevation MI within 3 days
2. Cardiogenic shock
3. Prior PCI within 1 year or any prior CABG anytime
4. Planned hybrid revascularization (PCI after CABG or CABG after PCI)
5. Planned single vessel revascularization (other than isolated left main disease)
6. Need for any cardiac surgical or interventional procedure other than coronary revascularization at the present time or anticipated within 3 years
7. Pregnancy (women of child-bearing potential must have a negative pregnancy test within 1 week before randomization) or intent to become pregnant within 1 year after randomization Unable to tolerate, obtain or comply with dual antiplatelet therapy for at least 3 months if presentation with stable CAD or 6 months if presentation with a troponin-positive acute coronary syndrome Current participation in another investigational drug or device study that has not reached its primary endpoint Life-expectancy less than 3 years due to concomitant non-cardiac conditions Any condition(s) are present that are likely to interfere with the study protocol procedures including medication adherence and follow-up through 10 years (e.g. mental disability, substance abuse, anticipated international relocation, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2033-03-15 (Estimated); Study Completion 2039-01-01 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite of all-cause death and time-averaged change from baseline in generic quality of life using the SF-12v2 | 5 years
  Generic quality of life (QOL) will be assessed by utilizing the 12-item Short Form Survey (SF-12v2). The score ranges from 1-100, with higher scores indicating a better health status. The win ratio will be used

SECONDARY OUTCOMES:
Time averaged change from baseline in disease-specific quality of life using the SAQ-OS | 5 years
  Disease-specific quality of life (QOL) will be assessed by utilizing the Seattle Angina Questionnaire overall summary (SAQ-OS) score. The score ranges from 1-100, with higher scores indicating a better health status.

OTHER OUTCOMES:
Time-averaged changes in PROMIS-29 Scores | 1 month, 3months, 6months, 12months and annually after procedure
  The PROMIS-29 instrument measures pain intensity on a scale of 0-10 plus 7 health domains: pain interference, fatigue, sleep disturbance, depressive symptoms, anxiety, physical function, and ability to participate in social roles. Each of the 7 domains is scored separately, with the lowest score for an individual domain being 4 and the highest being 20. Pain intensity is scored on the scale from 1-10. A mean of 50 and a standard deviation of 10 represent the general US population. A T-score rescales the raw scores to standardized scores. For most measures, higher T-scores indicate more of the concept being measured, except for physical function, which is reverse-scored (lower scores indicate worse function).
Time-averaged changes in EQ5D-VAS Scores | 1 month, 3months, 6months, 12months and annually after procedure
  The EQ5D-VAS records self-rated health status on a graduated visual analog scale (VAS) from 0-100, with higher scores for higher health-related quality of life. It also includes the EQ-5D descriptive system, which comprises 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Time-averaged changes in PHQ Scores | 1 month, 3months, 6months, 12months and annually after procedure
  The Patient Health Questionnaire (PHQ-8) is an 8-item questionnaire used to diagnose and quantify the severity of depressive symptoms. It is designed to evaluate the overall QOL of the individual and questions are based on the diagnostic criteria for Major Depressive Disorder outlined in the Diagnostic and Statistical Manual, 5th Edition (DSM-5). The lowest score is 0 and the highest score is 24. Scores ≥10 suggest a substantial burden of depressive symptoms.
Time-averaged changes in MoCA scores | 1 month, 3months, 6months, 12months and annually after procedure
  The telephone Montreal Cognitive Assessment (MoCA Blind or T-MoCA) is a tool to assess mild cognitive impairment. The MoCA BlindT-MoCA consists of 15 non-visual items that assesses different cognitive domains, including attention and concentration, memory, language, conceptual thinking, calculations, and orientation. The maximum score is 22 points with a score of 18 or below signifying mild cognitive dysfunction.
Number of days alive and out of hospital after procedure | up to 5 years after procedure
Time to death | 1 month after procedure
Time to death | 3 months after procedure
Time to death | 6 months after procedure
Time to death | 12 months after procedure
Time to death | 18 months after procedure
Time to death | 24 months after procedure
Time to death | 30 months after procedure
Time to death | 36 months after procedure
Time to death | 48 months after procedure
Time to death | 60 months after procedure
Time to death | 72 months after procedure
Time to death | 84 months after procedure
Time to death | 96 months after procedure
Time to death | 108 months after procedure
Time to death | 120 months after procedure
Time to cardiovascular death | 1 month after procedure
Time to cardiovascular death | 3 months after procedure
Time to cardiovascular death | 6 months after procedure
Time to cardiovascular death | 12 months after procedure
Time to cardiovascular death | 18 months after procedure
Time to cardiovascular death | 24 months after procedure
Time to cardiovascular death | 36 months after procedure
Time to cardiovascular death | 48 months after procedure
Time to cardiovascular death | 60 months after procedure
Time to cardiovascular death | 72 months after procedure
Time to cardiovascular death | 84 months after procedure
Time to cardiovascular death | 96 months after procedure
Time to cardiovascular death | 108 months after procedure
Time to cardiovascular death | 120 months after procedure
Time to non-cardiovascular death | 1 month after procedure
Time to non-cardiovascular death | 3 months after procedure
Time to non-cardiovascular death | 6 months after procedure
Time to non-cardiovascular death | 12 months after procedure
Time to non-cardiovascular death | 18 months after procedure
Time to non-cardiovascular death | 24 months after procedure
Time to non-cardiovascular death | 30 months after procedure
Time to non-cardiovascular death | 36 months after procedure
Time to non-cardiovascular death | 48 months after procedure
Time to non-cardiovascular death | 60 months after procedure
Time to non-cardiovascular death | 72 months after procedure
Time to non-cardiovascular death | 84 months after procedure
Time to non-cardiovascular death | 96 months after procedure
Time to non-cardiovascular death | 108 months after procedure
Time to non-cardiovascular death | 120 months after procedure
Time to myocardial infarction | 1 month after procedure
Time to myocardial infarction | 3 months after procedure
Time to myocardial infarction | 6 months after procedure
Time to myocardial infarction | 12 months after procedure
Time to myocardial infarction | 18 months after procedure
Time to myocardial infarction | 24 months after procedure
Time to myocardial infarction | 30 months after procedure
Time to myocardial infarction | 36 months after procedure
Time to myocardial infarction | 48 months after procedure
Time to myocardial infarction | 60 months after procedure
Time to myocardial infarction | 72 months after procedure
Time to myocardial infarction | 84 months after procedure
Time to myocardial infarction | 96 months after procedure
Time to myocardial infarction | 108 months after procedure
Time to myocardial infarction | 120 months after procedure
Time to stroke/transient ischemic attack | 1 month after procedure
Time to stroke/transient ischemic attack | 3 months after procedure
Time to stroke/transient ischemic attack | 6 months after procedure
Time to stroke/transient ischemic attack | 12 months after procedure
Time to stroke/transient ischemic attack | 18 months after procedure
Time to stroke/transient ischemic attack | 24 months after procedure
Time to stroke/transient ischemic attack | 30 months after procedure
Time to stroke/transient ischemic attack | 36 months after procedure
Time to stroke/transient ischemic attack | 48 months after procedure
Time to stroke/transient ischemic attack | 60 months after procedure
Time to stroke/transient ischemic attack | 72 months after procedure
Time to stroke/transient ischemic attack | 84 months after procedure
Time to stroke/transient ischemic attack | 96 months after procedure
Time to stroke/transient ischemic attack | 108 months after procedure
Time to stroke/transient ischemic attack | 120 months after procedure
Time to hospitalization | 1 month after procedure
Time to hospitalization | 3 months after procedure
Time to hospitalization | 6 months after procedure
Time to hospitalization | 12 months after procedure
Time to hospitalization | 18 months after procedure
Time to hospitalization | 24 months after procedure
Time to hospitalization | 30 months after procedure
Time to hospitalization | 36 months after procedure
Time to hospitalization | 48 months after procedure
Time to hospitalization | 60 months after procedure
Time to hospitalization | 72 months after procedure
Time to hospitalization | 84 months after procedure
Time to hospitalization | 96 months after procedure
Time to hospitalization | 108 months after procedure
Time to hospitalization | 120 months after procedure
Time to unplanned revascularization | 1 month after procedure
Time to unplanned revascularization | 3 months after procedure
Time to unplanned revascularization | 6 months after procedure
Time to unplanned revascularization | 12 months after procedure
Time to unplanned revascularization | 18 months after procedure
Time to unplanned revascularization | 24 months after procedure
Time to unplanned revascularization | 30 months after procedure
Time to unplanned revascularization | 36 months after procedure
Time to unplanned revascularization | 48 months after procedure
Time to unplanned revascularization | 60 months after procedure
Time to unplanned revascularization | 72 months after procedure
Time to unplanned revascularization | 84 months after procedure
Time to unplanned revascularization | 96 months after procedure
Time to unplanned revascularization | 108 months after procedure
Time to unplanned revascularization | 120 months after procedure
Time to atrial fibrillation/ atrial flutter | 1 month after procedure
Time to atrial fibrillation/ atrial flutter | 3 months after procedure
Time to atrial fibrillation/ atrial flutter | 6 months after procedure
Time to atrial fibrillation/ atrial flutter | 12 months after procedure
Time to atrial fibrillation/ atrial flutter | 18 months after procedure
Time to atrial fibrillation/ atrial flutter | 24 months after procedure
Time to atrial fibrillation/ atrial flutter | 30 months after procedure
Time to atrial fibrillation/ atrial flutter | 36 months after procedure
Time to atrial fibrillation/ atrial flutter | 48 months after procedure
Time to atrial fibrillation/ atrial flutter | 60 months after procedure
Time to atrial fibrillation/ atrial flutter | 72 months after procedure
Time to atrial fibrillation/ atrial flutter | 84 months after procedure
Time to atrial fibrillation/ atrial flutter | 96 months after procedure
Time to atrial fibrillation/ atrial flutter | 108 months after procedure
Time to atrial fibrillation/ atrial flutter | 120 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 1 month after procedure
Time to ventricular tachycardia/ventricular fibrillation | 3 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 6 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 12 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 18 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 24 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 30 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 36 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 48 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 60 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 72 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 84 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 96 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 108 months after procedure
Time to ventricular tachycardia/ventricular fibrillation | 120 months after procedure
Time to heart block | 1 month after procedure
Time to heart block | 3 months after procedure
Time to heart block | 6 months after procedure
Time to heart block | 12 months after procedure
Time to heart block | 18 months after procedure
Time to heart block | 24 months after procedure
Time to heart block | 30 months after procedure
Time to heart block | 36 months after procedure
Time to heart block | 48 months after procedure
Time to heart block | 60 months after procedure
Time to heart block | 72 months after procedure
Time to heart block | 84 months after procedure
Time to heart block | 96 months after procedure
Time to heart block | 108 months after procedure
Time to heart block | 120 months after procedure
Time to bleeding | 1 month after procedure
Time to bleeding | 3 months after procedure
Time to bleeding | 6 months after procedure
Time to bleeding | 12 months after procedure
Time to bleeding | 18 months after procedure
Time to bleeding | 24 months after procedure
Time to bleeding | 30 months after procedure
Time to bleeding | 36 months after procedure
Time to bleeding | 48 months after procedure
Time to bleeding | 60 months after procedure
Time to bleeding | 72 months after procedure
Time to bleeding | 84 months after procedure
Time to bleeding | 96 months after procedure
Time to bleeding | 108 months after procedure
Time to bleeding | 120 months after procedure
Time to vascular complications | 1 month after procedure
Time to vascular complications | 3 months after procedure
Time to vascular complications | 6 months after procedure
Time to vascular complications | 12 months after procedure
Time to vascular complications | 18 months after procedure
Time to vascular complications | 24 months after procedure
Time to vascular complications | 30 months after procedure
Time to vascular complications | 36 months after procedure
Time to vascular complications | 48 months after procedure
Time to vascular complications | 60 months after procedure
Time to vascular complications | 72 months after procedure
Time to vascular complications | 84 months after procedure
Time to vascular complications | 96 months after procedure
Time to vascular complications | 108 months after procedure
Time to vascular complications | 120 months after procedure
Time to heart failure | 1 month after procedure
Time to heart failure | 3 months after procedure
Time to heart failure | 6 months after procedure
Time to heart failure | 12 months after procedure
Time to heart failure | 18 months after procedure
Time to heart failure | 24 months after procedure
Time to heart failure | 30 months after procedure
Time to heart failure | 36 months after procedure
Time to heart failure | 48 months after procedure
Time to heart failure | 60 months after procedure
Time to heart failure | 72 months after procedure
Time to heart failure | 84 months after procedure
Time to heart failure | 96 months after procedure
Time to heart failure | 108 months after procedure
Time to heart failure | 120 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 1 month after procedure
Time to left ventricular assist device/orthotopic heart transplant | 3 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 6 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 12 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 18 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 24 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 30 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 36 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 48 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 60 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 72 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 84 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 96 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 108 months after procedure
Time to left ventricular assist device/orthotopic heart transplant | 120 months after procedure
Time to infection | 1 month after procedure
Time to infection | 3 months after procedure
Time to infection | 6 months after procedure
Time to infection | 12 months after procedure
Time to infection | 18 months after procedure
Time to infection | 24 months after procedure
Time to infection | 30 months after procedure
Time to infection | 36 months after procedure
Time to infection | 48 months after procedure
Time to infection | 60 months after procedure
Time to infection | 72 months after procedure
Time to infection | 84 months after procedure
Time to infection | 96 months after procedure
Time to infection | 108 months after procedure
Time to infection | 120 months after procedure
Time to acute kidney injury/chronic kidney disease | 1 month after procedure
Time to acute kidney injury/chronic kidney disease | 3 months after procedure
Time to acute kidney injury/chronic kidney disease | 6 months after procedure
Time to acute kidney injury/chronic kidney disease | 12 months after procedure
Time to acute kidney injury/chronic kidney disease | 18 months after procedure
Time to acute kidney injury/chronic kidney disease | 24 months after procedure
Time to acute kidney injury/chronic kidney disease | 30 months after procedure
Time to acute kidney injury/chronic kidney disease | 36 months after procedure
Time to acute kidney injury/chronic kidney disease | 48 months after procedure
Time to acute kidney injury/chronic kidney disease | 60 months after procedure
Time to acute kidney injury/chronic kidney disease | 72 months after procedure
Time to acute kidney injury/chronic kidney disease | 84 months after procedure
Time to acute kidney injury/chronic kidney disease | 96 months after procedure
Time to acute kidney injury/chronic kidney disease | 108 months after procedure
Time to acute kidney injury/chronic kidney disease | 120 months after procedure
Number of subjects with complete revascularization | 30 days after procedure
Number of subjects with reasonably complete revascularization | 30 days after procedure
Change in blood lipids | Baseline, 12 months post-procedure
Change in hemoglobin | Baseline, 12 months post-procedure
Change in LVEF | Baseline, 12 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mario Gaudino, MD, PhD, MSCE, FEBCTS, FACC, Principal Investigator — Weill Medical College of Cornell University; Gregg Stone, MD, FACC, MSCAI, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (18):
- United States (18):
  - Adventist Health Glendale, Glendale, California
  - Emory University, Atlanta, Georgia
  - Ascension St. Vincent Cardiovascular Research Institute, Carmel, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Englewood Hospital, Englewood, New Jersey
  - NewYork-Presbyterian Hospital - Queens, Flushing, New York
  - Icahn School of Medicine - Mount Sinai Morningside, New York, New York
  - Icahn School of Medicine - Mount Sinai Hospital, New York, New York
  - Columbia University Irving Medical Center/NewYork-Presbyterian Hospital, New York, New York
  - Weill Cornell Medicine/NewYork-Presbyterian Hospital, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Methodist Le Bonheur Healthcare, Memphis, Tennessee
  - Ascension Saint Thomas Hospital, Nashville, Tennessee
  - Baylor Scott and White, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No